CLINICAL TRIAL: NCT06881511
Title: Exploratory Study on the Efficacy of Betaine Hydrochloride in Treating Autoimmune Gastritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0911
Record Dates: First submitted 2025-03-12; First posted 2025-03-18 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Autoimmune Gastritis
Keywords: Autoimmune Gastritis; Iron-Deficiency Anemia; Stomach Neoplasms; Neuroendocrine Tumors; Betaine; Hydrochloride; Pepsin; Gastrointestinal Agents; Gastrins
MeSH Terms: conditions — Anemia, Iron-Deficiency; Stomach Neoplasms; Neuroendocrine Tumors | interventions — Control Groups; Betaine

STUDY DESIGN:
Intervention Model Description: This study will employ a linear mixed-effects model to analyze changes in primary outcomes (GSRS scores and serum gastrin levels), with the intervention effect evaluated through group-by-time interactions. For secondary outcomes, continuous variables will be analyzed using multiple linear regression, while categorical variables will be analyzed using logistic regression or Cox proportional hazards models. All models will adjust for baseline differences (via propensity score matching) and potential confounders. Model assumptions will be validated through residual analysis and diagnostic plots. Sensitivity analyses will include per-protocol vs intention-to-treat comparisons and alternative propensity score methods. Data analysis will be performed using R (version 4.0) or SAS (version 9.4).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: Observation Only (Control Group) (Other): Patients in this group will not receive any intervention and will only undergo regular follow-up and monitoring.
  Interventions: Other: No intervention (Control Group)
- Group B: Betaine Hydrochloride Supplementation (Experimental): Patients in this group will receive oral betaine hydrochloride (with pepsin) .
  Interventions: Dietary Supplement: Oral betaine hydrochloride (2 capsules, 3 times daily)

INTERVENTIONS:
Other: No intervention (Control Group) — Patients in this group will receive standard care and undergo regular follow-up and monitoring without any additional treatment.
  Arms: Group A: Observation Only (Control Group)
Dietary Supplement: Oral betaine hydrochloride (2 capsules, 3 times daily) — Oral betaine hydrochloride (with pepsin). Patients will take 2 capsules (648 mg per capsule) of betaine hydrochloride, 3 times daily with meals.
  Arms: Group B: Betaine Hydrochloride Supplementation

SUMMARY:
Autoimmune gastritis (AIG) is a chronic autoimmune disorder characterized by parietal cell destruction and oxyntic mucosal atrophy, leading to achlorhydria and intrinsic factor deficiency. These pathological changes impair iron and vitamin B12 absorption, resulting in iron-deficiency anemia, pernicious anemia, and neuropsychiatric manifestations. Notably, 4-12% of AIG patients develop type 1 gastric neuroendocrine tumors, while facing a 3-7 fold increased risk of gastric adenocarcinoma with an incidence of 0.9-9%.

Current management of AIG is limited to iron and vitamin B12 replacement, as no disease-modifying therapies exist. The progressive hypochlorhydria reduces pepsin activity, impairs gastric motility, and promotes small intestinal bacterial overgrowth (SIBO), causing dyspeptic symptoms and micronutrient malabsorption. Furthermore, gastric hypoacidity increases N-nitroso compound formation and triggers hypergastrinemia, elevating risks for both gastric cancer and neuroendocrine tumors.

This clinical trial investigates whether betaine hydrochloride (with pepsin) supplementation can restore gastric acidity and improve clinical outcomes in AIG. We will evaluate its effects on gastrin levels, gastrointestinal symptoms, exhaled gas markers (NO, H₂S, H₂, CH₄), anemia parameters, endoscopic atrophy scores, and incidence of gastric complications (hyperplastic polyps, neuroendocrine tumors, and adenocarcinoma). The study aims to provide evidence for a potential therapeutic strategy addressing both symptoms and long-term complications of AIG.

DETAILED DESCRIPTION:
Autoimmune gastritis (AIG) is a chronic progressive autoimmune disorder characterized by the destruction of gastric parietal cells, leading to atrophy of the acid-secreting gastric mucosa. The loss of parietal cells results in gastric acid deficiency and intrinsic factor deficiency, which in turn impairs the absorption of iron and vitamin B12, leading to clinical manifestations such as iron deficiency anemia, pernicious anemia, and neuropsychiatric symptoms. Studies indicate that 4-12% of AIG patients develop type 1 gastric neuroendocrine tumors (NETs), and these patients also face a 3-7 times higher risk of gastric adenocarcinoma, with an incidence rate ranging from 0.9% to 9%.

Currently, there are no anti-inflammatory, immunosuppressive, or biologic therapies available for AIG. Standard treatment involves iron and vitamin B12 supplementation. Due to progressive parietal cell destruction, AIG patients exhibit a hypochlorhydric state, which reduces pepsin activity, impairs gastric motility, and may lead to small intestinal bacterial overgrowth (SIBO), often causing symptoms such as dyspepsia. Additionally, low gastric acid levels can interfere with the absorption of trace elements like iron and calcium. Insufficient gastric acid also promotes bacterial overgrowth in the stomach and increases N-nitroso compounds, elevating the risk of gastric cancer. Furthermore, gastric hypochlorhydria triggers a feedback mechanism that stimulates gastrin secretion from antral G cells, resulting in hypergastrinemia, which increases the risk of neuroendocrine tumors. Supplementation with betaine hydrochloride (with pepsin) can lower gastric pH in AIG patients, restore gastric acidity, improve protein digestion, alleviate dyspeptic symptoms, enhance the absorption of vitamins and minerals, correct gastric dysbiosis and SIBO, and reduce the risk of gastric cancer and neuroendocrine tumors.

This study aims to evaluate the effects of betaine hydrochloride (with pepsin) on gastrin levels, gastrointestinal symptoms, exhaled gas markers (NO, H2S, H2, and CH4), iron deficiency anemia parameters, AIG atrophy scores, and the incidence of gastric complications (hyperplastic polyps, neuroendocrine tumors, and gastric cancer). The study is divided into two groups: Group A (follow-up only, serving as the control group) and Group B (oral betaine hydrochloride). The study adopts a non-randomized, open-label, parallel-controlled design, where participants choose either the experimental group (oral betaine) or the control group (follow-up only) based on their preference. Both groups will be followed in parallel, and outcome differences will be compared, supplemented by within-group pre- and post-intervention analyses.

The study population consists of AIG patients diagnosed at the Second Affiliated Hospital of Zhejiang University School of Medicine. The diagnostic criteria for AIG are based on our team's published article in Clinics and Research in Hepatology and Gastroenterology: "A real-world study on the characteristics of autoimmune gastritis: A single-center retrospective cohort in China." Inclusion criteria include: serum gastrin levels >300 pmol/L or a history of type 1 gastric NETs or early gastric cancer treated with endoscopic submucosal dissection (ESD), age between 18 and 80 years, and signed informed consent. Exclusion criteria include: allergy to betaine hydrochloride, presence of peptic ulcers, other conditions causing elevated gastrin levels, and refusal to sign informed consent.

Group A (control group) will undergo follow-up only without intervention, while Group B will receive oral betaine hydrochloride (2 capsules three times daily with meals). The primary outcomes include changes in serum gastrin levels and improvements in the Gastrointestinal Symptom Rating Scale (GSRS). Secondary outcomes include changes in iron deficiency anemia markers (serum iron, ferritin, hemoglobin), exhaled gas markers (NO, H2S, H2, CH4), AIG atrophy scores, and the incidence of gastric complications (hyperplastic polyps, NETs, and gastric cancer).

Data will be collected through questionnaires, laboratory tests, endoscopy, and pathological records, with propensity score matching (PSM) used to adjust for baseline differences. The study has been approved by the Ethics Committee of the Second Affiliated Hospital of Zhejiang University School of Medicine. Adverse events will be monitored regularly, and serious adverse events will be reported promptly to the ethics committee and regulatory authorities.

This study will provide critical evidence on the efficacy and safety of betaine hydrochloride in treating AIG, exploring a simple, cost-effective therapeutic approach to alleviate symptoms and reduce the risk of severe complications.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with autoimmune gastritis at the Second Affiliated Hospital of Zhejiang University School of Medicine, with the diagnostic criteria for autoimmune gastritis based on the article "A real-world study on the characteristics of autoimmune gastritis: A single-center retrospective cohort in China" published by our team in the journal Clinics and Research in Hepatology and Gastroenterology;
2. Gastrin levels greater than 300 pmol/L or a history of type 1 gastric neuroendocrine tumors or early gastric cancer treated with endoscopic submucosal dissection (ESD);
3. Age between 18 and 80 years;
4. Patients who have signed the informed consent form for the clinical trial.

Exclusion Criteria:

1. Patients allergic to betaine hydrochloride;
2. Patients with peptic ulcers;
3. Patients with any condition other than autoimmune gastritis that causes elevated gastrin levels (e.g., gastrinoma);
4. Patients who refuse to sign the informed consent form.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-03 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum Gastrin Levels | Baseline, 1 month, 3 months, 7 months, and 12 months.
  Comparison of the differences in serum gastrin levels before and after the trial within and between groups.
Gastrointestinal Symptom Scores | Baseline, 1 month, 3 months, 7 months, and 12 months.
  Gastrointestinal symptom scores will be assessed using the Gastrointestinal Symptom Rating Scale (GSRS) . Comparison of the differences in gastrointestinal symptom scores before and after the trial within and between groups.

SECONDARY OUTCOMES:
Exhaled Gas Markers (NO, H2S, H2, and CH4) | Baseline, 1 month, and 12 months.
  Comparison of the differences in exhaled gas marker levels (NO, H2S, H2, and CH4) before and after the trial within and between groups.
Iron Deficiency Anemia Indicators (Serum Iron, Ferritin, Hemoglobin) | Baseline, 1 month, and 12 months.
  Comparison of the differences in iron deficiency anemia indicators (serum iron, ferritin, and hemoglobin) before and after the trial within and between groups.
AIG Atrophy Score and Incidence of Gastric Complications | Baseline and 12 months.
  Comparison of the differences in AIG atrophy scores and the incidence of gastric complications (hyperplastic polyps, neuroendocrine tumors, and gastric cancer) before and after the trial within and between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Song M, Camargo MC, Katki HA, Weinstein SJ, Mannisto S, Albanes D, Surcel HM, Rabkin CS. Association of Antiparietal Cell and Anti-Intrinsic Factor Antibodies With Risk of Gastric Cancer. JAMA Oncol. 2022 Feb 1;8(2):268-274. doi: 10.1001/jamaoncol.2021.5395. PMID 34913949
- [Background] Rossi RE, Elvevi A, Sciola V, Mandarino FV, Danese S, Invernizzi P, Massironi S. Paradoxical association between dyspepsia and autoimmune chronic atrophic gastritis: Insights into mechanisms, pathophysiology, and treatment options. World J Gastroenterol. 2023 Jun 21;29(23):3733-3747. doi: 10.3748/wjg.v29.i23.3733. PMID 37398891
- [Background] Singh S, Chakole S, Agrawal S, Shetty N, Prasad R, Lohakare T, Wanjari M, Yelne S. A Comprehensive Review of Upper Gastrointestinal Symptom Management in Autoimmune Gastritis: Current Insights and Future Directions. Cureus. 2023 Aug 13;15(8):e43418. doi: 10.7759/cureus.43418. eCollection 2023 Aug. PMID 37706145
- [Background] Osmola M, Chapelle N, Vibet MA, Bigot-Corbel E, Masson D, Hemont C, Jirka A, Blin J, Tougeron D, Moussata D, Lamarque D, Josien R, Mosnier JF, Martin J, Matysiak-Budnik T. Iron and Vitamin B12 Deficiency in Patients with Autoimmune Gastritis and Helicobacter pylori Gastritis: Results from a Prospective Multicenter Study. Dig Dis. 2024;42(2):145-153. doi: 10.1159/000535206. Epub 2024 Jan 10. PMID 38198775
- [Background] Jove A, Lin C, Hwang JH, Balasubramanian V, Fernandez-Becker NQ, Huang RJ. Serum Gastrin Levels Are Associated With Prevalent Neuroendocrine Tumors in Autoimmune Metaplastic Atrophic Gastritis. Am J Gastroenterol. 2025 May 1;120(5):1140-1143. doi: 10.14309/ajg.0000000000003235. Epub 2024 Nov 26. PMID 39588964
- [Background] Chen C, Yang Y, Li P, Hu H. Incidence of Gastric Neoplasms Arising from Autoimmune Metaplastic Atrophic Gastritis: A Systematic Review and Case Reports. J Clin Med. 2023 Jan 30;12(3):1062. doi: 10.3390/jcm12031062. PMID 36769710
- [Background] Gomez Cifuentes JD, Sparkman J, Graham DY. Management of upper gastrointestinal symptoms in patients with autoimmune gastritis. Curr Opin Gastroenterol. 2022 Nov 1;38(6):600-606. doi: 10.1097/MOG.0000000000000878. Epub 2022 Sep 9. PMID 36165039
- [Background] Lenti MV, Rugge M, Lahner E, Miceli E, Toh BH, Genta RM, De Block C, Hershko C, Di Sabatino A. Autoimmune gastritis. Nat Rev Dis Primers. 2020 Jul 9;6(1):56. doi: 10.1038/s41572-020-0187-8. PMID 32647173
- [Background] Taylor L, McCaddon A, Wolffenbuttel BHR. Creating a Framework for Treating Autoimmune Gastritis-The Case for Replacing Lost Acid. Nutrients. 2024 Feb 27;16(5):662. doi: 10.3390/nu16050662. PMID 38474790
- [Background] Chen Y, Ji X, Zhao W, Lin J, Xie S, Xu J, Mao J. A real-world study on the characteristics of autoimmune gastritis: A single-center retrospective cohort in China. Clin Res Hepatol Gastroenterol. 2025 Apr;49(4):102556. doi: 10.1016/j.clinre.2025.102556. Epub 2025 Feb 15. PMID 39961485